CLINICAL TRIAL: NCT00578032
Title: Reconstructive Surgery For Head And Neck Cancer Patients: A Prospective Analysis Of Quality Of Life And Symptom Relief
Brief Title: Reconstructive Surgery For Head And Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-150; NCT00573625 (obsolete NCT alias)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Advanced Stage Head and Neck Cancer
Keywords: head; neck; cancer; reconstruction; quality of life; 07-150
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with head and neck malignancies that require simultaneous surgical resection and reconstruction of the ablative defect will be eligible to participate.
  Interventions: Behavioral: Quality of Life Questionaires & Interview: EORTC QLQ C-30, EORTC QLQ H&N-35, Health Behaviors, Subjective Significance Questionnaire, Qualitative Assessment

INTERVENTIONS:
Behavioral: Quality of Life Questionaires & Interview: EORTC QLQ C-30, EORTC QLQ H&N-35, Health Behaviors, Subjective Significance Questionnaire, Qualitative Assessment — All patients will complete the predefined questionnaires at the following four time points along the course of their care: preoperative clinic visit, and 3 months (±1 month), 6 months (±1), and 9 months (1 and +3) post-operatively. Completion of the questionnaires should take approximately 30 minutes

SUMMARY:
The goal of this study is to better understand the changes in symptoms and overall quality of life after head and neck surgery and reconstruction. "Quality of Life" means how you feel about your life as a result of your disease and its treatment. Learning about changes in patients' quality of life will help doctors and future patients make more informed treatment decisions.

DETAILED DESCRIPTION:
This prospective, longitudinal study will evaluate patient-reported quality of life and symptomatology immediately prior to and for up to one year following surgical resection and reconstruction head and neck malignancies.Patients with head and neck malignancies that require simultaneous surgical resection and reconstruction of the ablative defect will be eligible to participate.Quality of life and symptom relief will be evaluated by both domain and disease specific questionnaires at four time points: pre-operatively, and 3 months (±1 month), 6 months (±1), and 9 months (-1 and +3) post-operatively. These assessment points represent clinically significant events in patients' post-operative course following head and neck surgery. Studies have shown that quality of life decreases significantly at three months after surgery but then reapproaches baseline levels around one year (1). Pre-operative responses will serve as the baseline for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical resection and reconstruction for every stage head and neck malignancies at Memorial Sloan-Kettering Cancer Center.
* Patients at least 21 years of age

Exclusion Criteria:

* Patients who are less than 21 years old
* Patients who do not speak the English language
* Patients who are unable to comprehend the content of the questionnaires due to psychiatric disorders or cognitive impairment
* Patients who cannot complete the pre-operative questionnaires during consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and and neck malignancies hat require simultaneous surgical resection and reconstruction of the ablative defect will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
To describe overall pt-reported health-related QOL and cancer related symptoms pre-operatively and at 3, 6 and 9 mos following surgical resection and reconstruction for head & neck malignancies | 1 year

SECONDARY OUTCOMES:
To describe changes in patient-reported health-related quality of life and cancer-related symptoms within 9 or 12 months following surgical resection and reconstruction. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pusaic, MD, MHS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org